CLINICAL TRIAL: NCT04906057
Title: The Therapeutic Effects of Forced Aerobic Exercise in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Susan Linder, Assistant Staff, Physical Medicine and Rehabilitation, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1003
Record Dates: First submitted 2021-05-10; First posted 2021-05-28 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: aerobic exercise; gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: rater-blind, prospective randomized trial
Who Masked: Outcomes Assessor
Masking Description: Group allocation will be concealed to the individual obtaining all outcomes of interest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forced Aerobic Exercise (FE) (Experimental): The FE group (N=10) will complete 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's). The VE group (N=10) will exercise on an identical semi-recumbent cycle ergometer at their self-selected cadence without assistance.
  Interventions: Behavioral: Forced Aerobic Exercise (FE)
- Voluntary Aerobic Exercise (VE) (Active Comparator): The VE group (N=10) will exercise on an identical semi-recumbent cycle ergometer for 45 minutes at their self-selected cadence without assistance.
  Interventions: Behavioral: Voluntary Aerobic Exercise (VE)

INTERVENTIONS:
Behavioral: Forced Aerobic Exercise (FE) — High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
  Arms: Forced Aerobic Exercise (FE)
Behavioral: Voluntary Aerobic Exercise (VE) — Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometer
  Arms: Voluntary Aerobic Exercise (VE)

SUMMARY:
This project will investigate the feasibility and initial efficacy of two aerobic exercise training approaches, forced and voluntary, to improve motor function in persons with multiple sclerosis (MS). We hypothesize that intensive aerobic exercise training elicits a neurorepairative and neurorestorative response on the central nervous system, which may improve motor function as it relates to gait and mobility. Should aerobic cycling, forced or voluntary, improve gait and functional mobility in persons with MS, it would serve as a new model to restoring function, rather than current models that focus on compensation.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory and neurodegenerative disease of the central nervous system characterized by progressive loss of motor function, cognitive function, in addition to symptoms of fatigue and depression. These motor and non-motor symptoms negatively affect the individuals' walking ability, functional mobility, quality of life, ability to maintain gainful employment, and social engagement. Identifying rehabilitation approaches that may delay disease progression or restore lost neurologic function would have considerable impact in the field. The goal of this project is to investigate the feasibility and initial efficacy of forced or voluntary aerobic exercise training to improve gait, functional mobility, fatigue and quality of life in persons with multiple sclerosis (PwMS). Current rehabilitative approaches for PwMS focus on training compensatory strategies rather than restoring neurological function. Substantial evidence indicates that aerobic exercise (AE) training has the potential to enhance neurological function by restoring and repairing damaged cells, leading to improvements in gait, balance, and cognitive function in PwMS. Despite evidence of the potential disease-modifying properties of AE, numerous physical, behavioral, and logistical barriers prevent PwMS from achieving and maintaining AE of sufficient intensity and duration to capitalize on the neurophysiologic benefits of training. Forced exercise (FE) is a novel approach to AE training that has been successfully applied to individuals with Parkinson's disease and stroke, in which the voluntary efforts of the individual are augmented, allowing for disease-altering effects of intensive exercise training. During FE, pedaling cadence on a stationary cycle is augmented by a motor to assist, but not replace, the voluntary efforts of the individual. It is hypothesized that PwMS cannot sustain high rates of voluntary exercise necessary to elicit neural repair; therefore, FE is necessary to overcome physical, behavioral and logistical barriers to enhance neuroplasticity to improve gait, QOL, and the ability to participate in life activities. Positive results from our FE trials in Parkinson's disease and stroke have guided us in designing the scientific methodology for the proposed trial in PwMS. Twenty adults with relapsing-remitting MS and mild to moderate gait impairment will be randomized to undergo 1) FE or 2) voluntary aerobic exercise (VE). Both groups will attend 2X/week for 12 weeks. Exercise variables will be collected for each session as a measure of feasibility to determine how PwMS respond to each exercise approach. Clinical, biomechanical, and self-reported outcomes will be gathered prior to, after, and 4-weeks after the intervention to determine the effects of both modes of exercise on spatiotemporal and kinematic characteristics of gait, functional mobility, balance, fatigue, physical activity levels, and quality of life. Should our findings confirm our hypothesis that intensive exercise training can have disease-altering effects, a new direction for MS rehabilitation approaches would ensue, empowering PwMS to take control of their disease to improve function and reduce disability.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of RRMS with Expanded Disability Status Scale (EDSS) score between 1.5 and 6.5,
2. 18-75 years of age,
3. Deemed minimal risk for cardiovascular event using American College of Sports Medicine Exercise Pre-participation Criteria

Exclusion Criteria:

1. hospitalization for myocardial infarction, heart failure or heart surgery within 3 months,
2. serious cardiac arrhythmia,
3. hypertrophic cardiomyopathy,
4. severe aortic stenosis,
5. pulmonary embolus,
6. significant contractures,
7. dysphagia resulting in inability to sufficiently hydrate, and
8. other contraindication to exercise.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants identifying as male or female are eligible
Enrollment: 22 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Linder, DPT, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Forced Aerobic Exercise (FE): The FE group (N=11) completed 45 minutes of forced-rate aerobic exercise on a custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
- Voluntary Aerobic Exercise (VE): The VE group (N=7) completed aerobic exercise on an identical semi-recumbent cycle ergometer at their self-selected cadence without assistance for 45 minutes.
  Voluntary Aerobic Exercise (VE): Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometer
Period: Overall Study
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Aerobic Exercise (VE)
Started | 12 | 10
Completed | 11 | 7
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Forced Aerobic Exercise (FE): The FE group (N=11) completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
- Voluntary Aerobic Exercise (VE): The VE group (N=7) completed exercise on an identical semi-recumbent cycle ergometer for 45 minutes at their self-selected cadence without assistance.
  Voluntary Aerobic Exercise (VE): Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometer
- Total: Total of all reporting groups
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Aerobic Exercise (VE) | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants] — Population: 1. Participants withdrew due to unrelated injury
  2. Participants withdrew due to Covid-19
  1 Participant withdrew due to Covid-19
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 7 | 16
    >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1. Participants withdrew due to unrelated injury
  2. Participants withdrew due to Covid-19
  1 Participant withdrew due to Covid-19
  years | 53.6 (12.2) | 56.9 (7.9) | 54.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1. Participants withdrew due to unrelated injury
  2. Participants withdrew due to Covid-19
  1 Participant withdrew due to Covid-19
  Participants
    Female | 6 | 4 | 10
    Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1. Participants withdrew due to unrelated injury
  2. Participants withdrew due to Covid-19
  1 Participant withdrew due to Covid-19
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 10 | 7 | 17
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Exercise Duration
Description: Average exercise duration
Time Frame: collected during each exercise session (twice per week for 12 weeks)
Population: Completed participants in the FE & VE groups.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Forced Aerobic Exercise (FE): Results from this section include data from the Forced Exercise
  The FE group completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
- Voluntary Exercise (VE): The VE group completed exercises on an identical semi-recumbent cycle ergometer at their self-selected cadence without assistance for 45 minutes.
  Voluntary Aerobic Exercise (VE): Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometercle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise (VE)
Number analyzed (Participants) | 11 | 7
Minutes | 42.2 (2.4) | 42.2 (2.4)

2. Primary Outcome: Aerobic Intensity
Description: average percent max heart rate
Time Frame: Collected during each exercise session (twice per week for 12 weeks)
Population: FE + VE groups
Measure: Mean (Standard Deviation); unit: % Max HR
Groups:
- Forced Aerobic Exercise (FE): Results from this section include data from the Forced Exercise group.
  The FE group completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise (VE)
Number analyzed (Participants) | 11 | 7
% Max HR | 0.63 (0.07) | .70 (0.05)

3. Primary Outcome: Exercise Cadence
Description: Average Exercise Cadence (cycling rate)
Time Frame: collected during each exercise session (twice per week for 12 weeks)
Population: Completed participants within the FE & VE groups
Measure: Mean (Standard Deviation); unit: revolutions per minute
Groups:
- Forced Aerobic Exercise (FE): Results from this section includes data the Forced Exercise.
  The FE group completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise (VE)
Number analyzed (Participants) | 11 | 7
revolutions per minute | 69.1 (11.1) | 64.5 (16.7)

4. Primary Outcome: Six Minute Walk Test
Description: The distance walked over 6 minutes is measured on an oval walking track
Time Frame: Week 0 (baseline), Week 13 (post exercise sessions)
Population: Week (0) Baseline + EOT Week (13)
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Forced Aerobic Exercise (FE): The FE group completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
- Voluntary Exercise: The VE group completed exercises on an identical semi-recumbent cycle ergometer at their self-selected cadence without assistance for 45 minutes.
  Voluntary Aerobic Exercise (VE): Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise
Number analyzed (Participants) | 11 | 7
Meters
  Baseline | 339.1 (123.3) | 345.9 (110.7)
  EOT | 338.3 (111.5) | 373.6 (128.6)

5. Primary Outcome: Gait Velocity
Description: Spatio-temporal and kinematic parameters of gait will be obtained using 3-D motion capture and an instrumented walkway.
Time Frame: Week 0 (baseline), Week 13 (post exercise sessions)
Population: Data was obtained using a ZENO & Caren walking pad; however, one participant was unable to complete this outcome measure due to unsteady gait.
Measure: Mean (Standard Deviation); unit: Meters per second
Groups:
- Forced Aerobic Exercise (FE): Results from this section includes data from both the Forced Exercise and the Voluntary Exercise Group.
  The FE group completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise
Number analyzed (Participants) | 10 | 7
Meters per second
  Zeno Velocity Self-Paced Baseline (average) | 90.6 (17.3) | 91.5 (30.6)
  Zeno Velocity Fast-Paced Baseline (average) | 122.4 (19.3) | 131.0 (13.0)
  CAREN Walking Speed Baseline (Average) | 0.54 (.28) | 0.65 (0.30)

6. Primary Outcome: PROMIS-29
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in the general population and with individuals living with chronic conditions. Raw scores were converted to T-scores (using an adult referent population) ranging from 0-100 with a mean of 50 and standard deviation (SD) of 10 in the referent population. For the PROMIS-29 symptom-related domains (anxiety, depression, fatigue, sleep disturbance, and pain interference), higher scores represent greater symptom burden (worse function). For the physical and participation domains, higher scores represent greater levels of function. Pain intensity is scored separately using a 0-10 scaler with higher scores representing greater pain.
Time Frame: Week 0 (baseline), Week 13 (post exercise sessions)
Population: Each participant completed the PROMIS-29 assessment at baseline. Some participants chose not to complete the EOT questionnaire, hence the overall number of participants for the EOT testing is fewer than the baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Forced Aerobic Exercise (FE) + Voluntary Exercise (VE): Results from this section includes data from both the Forced Exercise and the Voluntary Exercise Group.
  The FE group completed 45 minutes of FE on the custom-engineered cycle designed to augment pedaling rate to greater than 70 revolutions per minute (RPM's).
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) + Voluntary Exercise (VE) | Voluntary Exercise
Number analyzed (Participants) | 11 | 7
Units on a scale
  PROMIS Physical at baseline | 40.2 (7.8) | 40.8 (7.8)
  PROMIS Physical at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Physical at EOT | 40.0 (6.0) | 40.0 (5.0)
  PROMIS Anxiety at baseline | 46.6 (7.6) | 49.5 (12.3)
  PROMIS Anxiety at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Anxiety at EOT | 45.8 (6.3) | 45.6 (7.3)
  PROMIS Depression at baseline | 46.1 (7.8) | 46.5 (10.8)
  PROMIS Depression at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Depression at EOT | 45.7 (7.7) | 45.8 (6.6)
  PROMIS Fatigue at baseline | 50.8 (11.5) | 53.5 (5.2)
  PROMIS Fatigue at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Fatigue at EOT | 48.6 (11.0) | 47.9 (3.3)
  PROMIS Sleep Disturbance at baseline | 43.2 (5.4) | 45.8 (9.8)
  PROMIS Sleep Disturbance at EOT | 42.9 (6.1) | 44.9 (7.8)
  PROMIS Participation at baseline | 50.5 (7.0) | 49.2 (7.9)
  PROMIS Participation at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Participation at EOT | 53.6 (8.8) | 52.0 (8.1)
  PROMIS Pain Interference at baseline | 52.7 (10.4) | 54.9 (7.2)
  PROMIS Pain Interference at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Pain Interference at EOT | 46.5 (8.2) | 50.1 (7.7)
  PROMIS Pain Intensity at baseline | 3.5 (2.7) | 4.1 (1.6)
  PROMIS Pain Intensity at EOT: number analyzed (Participants) | 10 | 5
  PROMIS Pain Intensity at EOT | 2.6 (1.8) | 3.2 (1.9)

7. Primary Outcome: Modified Fatigue Impact Scale (MFIS)
Description: The MFIS is a 21-item self-reported measure of how fatigue impacts the lives of persons with multiple sclerosis. This instrument provides an assessment of the effects of fatigue as it relates to physical, cognitive, and psychosocial functioning. Participants rate on a 5-point Likert scale, with 0 = 'Never' to 4 = 'Almost always' their agreement with 21 statements. Total score (0-84) and subscales for physical (0-36), cognitive (0-40) and psychosocial functioning (0-8). Higher numbers indicate greater fatigue in all domains.
Time Frame: Week 0 (baseline), Week 13 (post exercise sessions)
Population: Each participant completed the Modified Fatigue Impact Scale (MFIS) assessment at baseline. Some participants chose not to complete the EOT questionnaire, hence the overall number of participants for the EOT testing is fewer than the baseline.
Measure: Mean (Standard Deviation); unit: score on Likert scale
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise
Number analyzed (Participants) | 11 | 7
score on Likert scale
  MFIS total score at baseline | 21.9 (18.5) | 33.4 (12.8)
  MFIS total score at EOT: number analyzed (Participants) | 10 | 5
  MFIS total score at EOT | 18.6 (18.7) | 20.2 (7.5)
  MFIS Physical Subscale at baseline | 14.0 (10.6) | 18.7 (6.9)
  MFIS Physical Subscale at EOT: number analyzed (Participants) | 10 | 5
  MFIS Physical Subscale at EOT | 9.9 (10.3) | 11.8 (3.6)
  MFIS Cognitive Subscale at baseline | 7.6 (7.4) | 12.3 (7.3)
  MFIS Cognitive Subscale at EOT: number analyzed (Participants) | 10 | 5
  MFIS Cognitive Subscale at EOT | 7.2 (6.9) | 6.8 (6.6)
  MFIS Psychosocial Subscale at baseline | 2.0 (1.90) | 2.3 (2.1)
  MFIS Psychosocial Subscale at EOT: number analyzed (Participants) | 10 | 5
  MFIS Psychosocial Subscale at EOT | 1.5 (1.7) | 1.6 (1.7)

8. Primary Outcome: Multiple Sclerosis Manual Dexterity Test
Description: Assessment examining cognitive and hand function for persons with MS
Time Frame: Week 0 (baseline), Week 13 (post exercise sessions)
Population: One forced exercise participant was unable to complete the Manual Dexterity test on the left side at baseline.
Measure: Mean (Standard Deviation); unit: Time in Seconds
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise (VE)
Number analyzed (Participants) | 11 | 7
Time in Seconds
  Manual Dexterity Test (Right) at baseline | 31.4 (8.2) | 24.3 (4.1)
  Manual Dexterity Test (right) at EOT | 32.4 (7.8) | 23.9 (4.4)
  Manual Dexterity Test (Left) at baseline: number analyzed (Participants) | 11 | 6
  Manual Dexterity Test (Left) at baseline | 33.8 (5.8) | 25.4 (2.0)
  Manual Dexterity Test (left) at EOT | 35.4 (9.8) | 39.6 (35.9)

9. Primary Outcome: Processing Speed Test
Description: Assessment examining processing speed using an tablet-based measure developed to closely resemble the symbol digit modalities test. Participants match symbols to digits over a 2-minute trial. The number of correct matches represents the score, with higher correct matches indicative of better processing speed performance. The low range of possible scoring is 0 with no upper range limit. In a study by Rao and colleagues (2017), persons with MS scored and average of 51.1 (+/- 11.9) on the first trial and 52.8 (+/- 2.0) on the second trial. One trial was conducted in this study.
Time Frame: Week 0 (baseline), Week 13 (post exercise sessions)
Population: One participant from the VE group could not complete the processing speed test.
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Exercise
Number analyzed (Participants) | 10 | 7
number correct
  Processing speed test total correct at baseline | 43.0 (8.0) | 55.3 (8.5)
  Processing speed test total correct at EOT | 45.1 (9.4) | 57.4 (9.8)

10. Secondary Outcome: To Investigate the Role of Klotho in Promoting Neuroprotection.
Description: Laboratory Assessment: Blood draws will be conducted at 4 different points in time to determine the acute and long-term change in serum Klotho; at week one session one, pre- and post-exercise, and at the last session12-week exercise intervention, pre- and post-exercise.
Time Frame: Week 1 (exercise session 1), Week 12 (exercise session 24)
Population: Participants in this data set have completed the entire 12 weeks of the prescribed exercise session.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Voluntary Aerobic Exercise (VE): The VE group completed exercises on an identical semi-recumbent cycle ergometer at their self-selected cadence without assistance for 45 minutes.
  Voluntary Aerobic Exercise (VE): Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Aerobic Exercise (VE)
Number analyzed (Participants) | 12 | 6
pg/mL
  Klotho (Baseline Pre-Exercise): number analyzed (Participants) | 12 | 5
  Klotho (Baseline Pre-Exercise) | 1273.3 (787.7) | 1100.4 (878.0)
  Klotho (Baseline Post-Exercise): number analyzed (Participants) | 12 | 5
  Klotho (Baseline Post-Exercise) | 929.5 (661.1) | 1166.4 (745.4)
  Klotho (Final Session pre-exercise): number analyzed (Participants) | 12 | 5
  Klotho (Final Session pre-exercise) | 948.3 (550.2) | 1019.4 (608.7)
  Klotho (Final Session post-exercise): number analyzed (Participants) | 12 | 5
  Klotho (Final Session post-exercise) | 1265.8 (940.2) | 154.4 (1104.1)
  Neurofilament light (Baseline) | 14.6 (7.5) | 14.5 (7.3)
  Neurofilament light (Final Session) | 16.5 (6.4) | 15.0 (4.0)

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected up to 19 weeks from start to completion of the study.
Groups:
- Forced Aerobic Exercise (FE): This section includes data from all randomized participants in the forced exercise group
  The FE group (N=12) completed 45 minutes of FE on the custom-engineered cycle designed to augment the pedaling rate to greater than 70 revolutions per minute (RPM's). The VE group (N=10) will exercise on an identical semi-recumbent cycle ergometer at their self-selected cadence without assistance.
  Forced Aerobic Exercise (FE): High-rate aerobic exercise on a semi-recumbent custom-designed stationary cycle ergometer
- Voluntary Aerobic Exercise (VE): This section includes data from all randomized participants in the the voluntary exercise group
  The VE group (N=10) completed the exercise on an identical semi-recumbent cycle ergometer for 45 minutes at their self-selected cadence without assistance.
  Voluntary Aerobic Exercise (VE): Voluntary-rate aerobic exercise on a semi-recumbent stationary cycle ergometer
Arm/Group | Forced Aerobic Exercise (FE) | Voluntary Aerobic Exercise (VE)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/10
Other Adverse Events (participants affected / at risk) | 2/12 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forced Aerobic Exercise (FE) (N=12) | Voluntary Aerobic Exercise (VE) (N=10)
STEMI (Cardiac disorders) | 1 (1) | 0 (0) — Heart attack
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forced Aerobic Exercise (FE) (N=12) | Voluntary Aerobic Exercise (VE) (N=10)
Covid-19 Diagnosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04906057/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04906057/SAP_001.pdf